CLINICAL TRIAL: NCT00438321
Title: Effect of Increasing Testosterone on Insulin Sensitivity in Men With the Metabolic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI relocated
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); American Diabetes Association (Other)
Responsible Party: Principal Investigator, Frances Hayes, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-001526
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Syndrome
Keywords: Overweight; obesity; testosterone; diabetes; metabolic syndrome; aging
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Diabetes Mellitus | interventions — Goserelin; Testosterone; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo injection, gel and pill
  Interventions: Other: Placebo
- Testosterone only (Active Comparator): Zoladex 3.6 mg IM injection Testosterone 7.5 g gel (AndroGel) transdermally daily Anastrozole 10 mg (Arimidex) orally daily
  Interventions: Drug: Zoladex; Drug: Testosterone gel; Drug: Anastrozole Pill
- Testosterone and Estrogen (Active Comparator): Zoladex 3.6 mg IM injection Testosterone 7.5 g gel (AndroGel) transdermally Placebo pill orally daily
  Interventions: Drug: Zoladex; Drug: Testosterone gel

INTERVENTIONS:
Drug: Zoladex
  Arms: Testosterone and Estrogen; Testosterone only
Drug: Testosterone gel
  Other Names: AndroGel
  Arms: Testosterone and Estrogen; Testosterone only
Drug: Anastrozole Pill
  Other Names: Arimidex
  Arms: Testosterone only
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the effect of testosterone treatment on insulin in men with the metabolic syndrome with testosterone levels at or below the lower end of the normal range.

DETAILED DESCRIPTION:
The metabolic syndrome is a medical condition defined by high cholesterol levels, high blood pressure, increased abdominal obesity (gain in fat around the region of the stomach), and insulin resistance. Insulin is the hormone that your body produces to decrease the levels of sugar in your blood. A person that is insulin resistant needs more insulin to decrease blood sugar levels than a normal person does. Insulin resistance can lead to type 2 diabetes, which is one of the most common illnesses in the United States.

There is evidence pointing to a relationship between insulin and testosterone in men (testosterone is the male sex hormone that is produced in the testes). As men get older their testosterone levels decrease while their weight and insulin resistance tends to increase. The purpose of this research study is to learn more about the details of the relationship between insulin and testosterone. A clearer understanding of this relationship can have an important impact on public health due to the high rate of health problems associated with diabetes, obesity, and heart disease.

We are looking for men between the ages of 50-75 with the metabolic syndrome to participate in this research study. Participation in this study involves taking medication and/or placebo (a placebo looks exactly like the study medication but contains no active drug), blood tests, muscle biopsies, and imaging scans. This study involves outpatient visits. Subjects are paid up to $500 for completing the study.

ELIGIBILITY:
Inclusion Criteria:

Stable weight for previous three months (no weight change greater than or equal to +/-10 lbs)

Exclusion Criteria:

* No new diagnosis of type 2 diabetes or on oral hypoglycemic agents
* No history of testicular disorders
* No history of bleeding disorders (i.e. Pulmonary Embolism, Deep Vein Thrombosis, stroke, hypercoagulable syndrome)
* No history of prostate cancer
* No previous diagnosis of osteoporosis
* No history of sleep apnea (subjects will also be excluded if at their baseline assessment they admit to heavy snoring, restless sleep, and/or excessive daytime somnolence)
* No symptoms of urinary outflow obstruction or medications for prostate disease
* No illicit drug use or heavy alcohol use (>4 drinks/day)

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02-26 (Actual); Study Completion 2010-02-26 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 3 months
  Assessed by euglycemic-hyperinsulinemic clamp

SECONDARY OUTCOMES:
Resting energy expenditure | 3 months
  Indirect calorimetry
Lipid profile | 3 months
  Fasting lipids
Body composition | 3 months
  DXA scan
Intramyocellular fat | 3 months
  MR spectroscoopy

CONTACTS AND LOCATIONS:
Overall Officials: Frances J Hayes, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pitteloud N, Hardin M, Dwyer AA, Valassi E, Yialamas M, Elahi D, Hayes FJ. Increasing insulin resistance is associated with a decrease in Leydig cell testosterone secretion in men. J Clin Endocrinol Metab. 2005 May;90(5):2636-41. doi: 10.1210/jc.2004-2190. Epub 2005 Feb 15. PMID 15713702
- [Background] Pitteloud N, Mootha VK, Dwyer AA, Hardin M, Lee H, Eriksson KF, Tripathy D, Yialamas M, Groop L, Elahi D, Hayes FJ. Relationship between testosterone levels, insulin sensitivity, and mitochondrial function in men. Diabetes Care. 2005 Jul;28(7):1636-42. doi: 10.2337/diacare.28.7.1636. PMID 15983313
- See also: Related Info — http://www.massgeneral.org/reproendo/pages/reu_study_subject.htm